CLINICAL TRIAL: NCT03134326
Title: Rainbow R2-25 vs. R1-25 SpHb Sub-Range Performance Equivalence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: TR18735-1029
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test group (Experimental): All subjects will be enrolled in the test group and will receive both R1-25 and R2-25 Pulse Oximeter Sensors
  Interventions: Device: R1-25 and R2-25 Pulse Oximeter Sensor

INTERVENTIONS:
Device: R1-25 and R2-25 Pulse Oximeter Sensor

SUMMARY:
In this study, the concentration of hemoglobin was measured using noninvasive pulse oximeter sensors and compared against the hemoglobin measurement from the subject's blood sample under controlled conditions. Data collected in the study was in the sub-range of 12-17 g/dL in the device's 8-17 g/dL specification range.

The purpose of the study was to evaluate a change in the sensor component and to assess performance equivalence in the sub-range. The performance of non-invasive hemoglobin is not uniform across the accuracy range.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Healthy

Exclusion criteria:

* Do not understand the study and the risks involved
* Deemed ineligible by study test personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-06-18 (Actual); Primary Completion 2009-07-02 (Actual); Study Completion 2009-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Group
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Sub-Range Performance Equivalence of R2-25 and R1-25 Sensors by ARMS Calculation
Description: Sub-range performance equivalence was determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter sensor to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square (Arms) error value. In order to obtain the Arms value, the blood sample hemoglobin value is subtracted from the pulse oximeter hemoglobin value for a number of samples, the average of this difference is computed as the bias. The standard deviation of these differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours
Measure: Number; unit: g/dL
Arm/Group | Test Group
Number analyzed (Participants) | 21
g/dL
  R2-25 sensor | 1.33
  R1-25 sensor | 1.41

ADVERSE EVENTS:
Arm/Group | Test Group
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less